CLINICAL TRIAL: NCT01167543
Title: Relationship and Pathophysiology of Gastroesophageal Reflux and Dental/Periodontal Disease
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Melvin B. Heyman MD MPH, University of California, San Francisco
Other Study IDs: MA-L-017
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-05

CONDITIONS: Gastroesophageal Reflux; Dental Erosion
MeSH Terms: conditions — Gastroesophageal Reflux; Tooth Erosion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pediatric patients with symptoms or diagnosis of GER
- Control group of pediatric subjects with no symptoms of GER.

SUMMARY:
This study investigates the prevalence and pathophysiology of dental and periodontal involvement in pediatric patients with symptomatic or asymptomatic gastroesophageal reflux (GER) or gastroesophageal reflux disease (GERD). Primary objectives are to compare the prevalence of oral disease in children with and without a diagnosis or symptoms/signs of GERD in a cross-sectional study. Secondary objectives are to examine factors that might lead to the pathogenesis of the dental and periodontal lesions observed in this group of subjects.

The primary hypothesis is to prove that children aged 10-18 years diagnosed with or having symptoms or signs of GERD have a significantly higher amount of dental erosions in comparison to a matched control group.

Secondary hypotheses are that children aged 10 - 18 years diagnosed with or having signs of GER have higher DMFS (Decayed, Missing, Filled permanent tooth Surfaces) rates, higher SBI (Sulcus Bleeding Index) rates, worse Periodontal status, and lower saliva buffering capacity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 9.0 to 18.0 years, of either gender
* Able to give verbal / written assent / consent themselves and/or informed consent from a parent/guardian
* Willing to comply with all study procedures and protocols,
* Willing to get dental photographs and impressions taken
* Willing to sign the "Authorization for Release of Personal Health Information and Use of Personally Unidentified Study Data for Research" form

Exclusion Criteria:

* Subjects suffering from systemic diseases, significant past or medical history with conditions that may affect oral health or oral flora (i.e. diabetes, HIV, heart conditions that require antibiotic prophylaxis)
* Other conditions that may decrease the likelihood of adhering to study protocol,
* Subjects who will leave the area and are unable to complete the study.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric Specialty Clinics and General Pediatric Clinics at the University of California, San Francisco
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2005-09; Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco Dental School, San Francisco, California, United States